CLINICAL TRIAL: NCT06871111
Title: The Microbiota Augmentation to Reestablish Commensal Organisms (MARCO) Trial
Acronym: MARCO
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB24-0560
Record Dates: First submitted 2025-02-13; First posted 2025-03-11 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-08

CONDITIONS: Liver Diseases; Liver Failure; Cirrhosis, Liver
MeSH Terms: conditions — Liver Diseases; Liver Failure; Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: Using adaptive trial design, there is the potential that patients could receive 1 of 9 different 8-member bacterial consortia. After the initial 8 subjects complete treatment with Consortium A, fecal metagenomic and metabolomic information will be used to classify results into 1 of 5 different conditions (Condition 1, 2(i), 2(ii), 2(iii), or 3). The subsequent 16 subjects will be given consortium based on these results. If Consortium A has good engraftment and metabolite production, the following 16 subjects will also be given Consortium A. Otherwise, patients will be given two sub-consortia (B-E), and subjects will be randomized 1:1 into the two sub-consortia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Commensal Consortium A (Experimental): Stage 1: 1st 8 patients enrolled will receive Consortium A. This consortium contains 7 different organisms.
  Interventions: Biological: Commensal Bacteria Strains
- Commensal Consortium B1 (Experimental): Stage 2: Based on fecal metagenomic and metabolomic data from Stage 1, subjects may be assigned to this Commensal Consortium. This consortium contains 7 different organisms.
  Interventions: Biological: Commensal Bacteria Strains
- Commensal Consortium B2 (Experimental): Stage 2: Based on fecal metagenomic and metabolomic data from Stage 1, subjects may be assigned to this Commensal Consortium. This consortium contains 7 different organisms.
  Interventions: Biological: Commensal Bacteria Strains
- Commensal Consortium C1 (Experimental): Stage 2: Based on fecal metagenomic and metabolomic data from Stage 1, subjects may be assigned to this Commensal Consortium. This consortium contains 7 different organisms.
  Interventions: Biological: Commensal Bacteria Strains
- Commensal Consortium C2 (Experimental): Stage 2: Based on fecal metagenomic and metabolomic data from Stage 1, subjects may be assigned to this Commensal Consortium. This consortium contains 7 different organisms.
  Interventions: Biological: Commensal Bacteria Strains
- Commensal Consortium D1 (Experimental): Stage 2: Based on fecal metagenomic and metabolomic data from Stage 1, subjects may be assigned to this Commensal Consortium. This consortium contains 7 different organisms.
  Interventions: Biological: Commensal Bacteria Strains
- Commensal Consortium D2 (Experimental): Stage 2: Based on fecal metagenomic and metabolomic data from Stage 1, subjects may be assigned to this Commensal Consortium. This consortium contains 8 different organisms.
  Interventions: Biological: Commensal Bacteria Strains
- Commensal Consortium E1 (Experimental): Stage 2: Based on fecal metagenomic and metabolomic data from Stage 1, subjects may be assigned to this Commensal Consortium. This consortium contains 7 different organisms.
  Interventions: Biological: Commensal Bacteria Strains
- Commensal Consortium E2 (Experimental): Stage 2: Based on fecal metagenomic and metabolomic data from Stage 1, subjects may be assigned to this Commensal Consortium. This consortium contains 7 different organisms.
  Interventions: Biological: Commensal Bacteria Strains

INTERVENTIONS:
Biological: Commensal Bacteria Strains — 7 doses containing 7 capsules will be administered over 7-10 days
  Other Names: Lyophilized live commensal bacterial strains (Live Biotherapeutic Product); Commensal Consortium

SUMMARY:
The Microbiota Augmentation to Reestablish Commensal Organisms (MARCO) trial is a single center prospective adaptive phase 1b clinical trial in patients who are hospitalized with complications of liver disease and have low fecal metabolite levels (butyrate and deoxycholic acid). The study intervention is 1 of 9 novel live Commensal Consortia each containing eight commensal bacterial strains derived from healthy donors. The primary objective of the study is to determine safety and tolerability of Commensal Consortia administration.

DETAILED DESCRIPTION:
The global burden of chronic liver disease (CLD) continues to rise. CLD is often clinically silent until an initial decompensation event, after which care is largely supportive without the ability to significantly modify the underlying disease with current therapies. Due to the high rates of infection in patients with liver disease, empiric, broad spectrum antibiotics are commonly prescribed. This practice is associated with altered gut microbiome compositions, reduced levels of health-promoting bacterial metabolites and high levels of antibiotic resistant organisms, findings that correlate with poor clinical outcomes including infection, repeat hepatic decompensation, re-hospitalization and death.

The primary objective of this clinical trial is to test the safety of commensal bacterial strain combinations designed to reconstitute microbiota compositions and metabolite production in patients with liver disease and profound dysbiosis as measured by low fecal metabolite (butyrate and deoxycholic acid) concentrations. The exploratory outcomes include strain engraftment and bacterial metabolite production.

The trial will occur in two phases. During the first phase, 8 patients will be recruited and administered the same combination of bacterial strains for 7 doses. Patients will be monitored for safety and tolerability. Additionally, fecal samples will be collected to assess for the presence of administered strains and fecal metabolite production.

After the first phase, additional combinations of bacteria will be chosen based upon the safety, engraftment and metabolite production in the first phase. In this adaptive phase, an additional 16 subjects will be enrolled and randomized to one of two additional consortia. In the two phases, a total of 24 patients will be enrolled, and each will be followed for 12 months to assess both primary (safety and tolerability) and exploratory (engraftment and metabolite production) outcomes. The investigators anticipate completing enrollment within 12 months of trial initiation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of liver disease, liver failure, and/or cirrhosis
* All patients will be hospitalized and have a hepatology consult in place.
* They will be identified as having liver disease, liver failure, and/or cirrhosis based on a combination of at least one of the following:

  * Labs demonstrating elevated liver chemistries (AST and ALT), elevated serum bilirubin levels, prolonged INR, or radiologic evidence of cirrhosis (e.g. nodular liver contour);
  * Liver biopsy results; and/or
  * Clinical or radiologic evidence of portal hypertension (e.g. splenomegaly, known varices, ascites, or hepatic venous pressure gradient ≥ 10mmHg).
  * All diagnoses will be confirmed by the attending hepatologist's interpretation and consult note attestation.
* Admitted to the hospital for hepatic decompensation
* MELD score ≤ 30 at time of enrollment
* Subject has ≤ 700µM butyrate and ≤ 10µM deoxycholate in fecal sample

Exclusion Criteria:

* MELD score >30 at time of enrollment
* Patients receiving any antibiotics for treatment of an infection.
* Chronic or prophylactic antibiotic administration other than rifaximin, ciprofloxacin, or trimethoprim-sulfamethoxazole.

  -Rifaximin will be either temporarily held or switched to another non-antibiotic therapy (e.g. lactulose or sodium benzoate) during the treatment phase of the trial. Potential subjects in whom the treating hepatologist deem it unsafe to pause or switch from Rifaximin therapy during the 7-10 day treatment phase will be excluded from the study.
* Patients who are currently admitted to the intensive care unit for vasoactive support or mechanical ventilation.
* Patients meeting the North American Consortia for Study of End Stage Liver Disease (NACSELD) criteria for acute-on-chronic liver failure (ACLF) with ≥ 2 organ failures by NACSELD-ACLF criteria at time of enrollment.
* Patients with known intestinal barrier dysfunction, including active GI bleeding, enteropathy (including celiac disease), clinically active inflammatory bowel disease (Crohn's or Ulcerative Colitis), ischemic colitis, microscopic colitis, graft versus host disease (GVHD), or gastrointestinal malignancy.

  o Active inflammatory bowel disease (IBD) will be defined based on a combination of:
  * Symptoms (diarrhea and/or abdominal pain without another explanation)
  * Laboratory evidence of inflammation (e.g. elevated CRP or fecal calprotectin without another explanation); and
  * Either radiologic, endoscopic, and/or histologic evidence of active IBD.
  * If IBD is suspected, this will be investigated with the general GI consult service prior to approaching for enrollment.
  * If patients carry a diagnosis of IBD but do not meet the above criteria, they will be eligible for enrollment unless their IBD is managed with a systemic immunosuppression medication (e.g. anti-TNF-alpha therapy).
  * If any form of the above intestinal disorders is suspected, they will be investigated with the general GI consult service prior to approaching for enrollment.
* Profoundly immunocompromised patients, including patients with primary immunodeficiency, solid organ transplant recipients, any history of hematopoietic stem cell transplant (HSCT), ongoing cancer treatment, neutropenia < 500 cells/mm3, HIV untreated or with CD4 < 200 cells/mm3, immunosuppressive medications, including rituximab, anti-cytokine therapy, anti-rejection medications, chronic corticosteroids (a dose ≥ 20mg of prednisone daily for ≥ 1 month), biologic therapy for autoimmune condition.
* Patients with delayed gastrointestinal motility as evidenced by ≤ 2 bowel movements per week at the time of enrollment.
* Patients who are allergic to both ampicillin/sulbactam and meropenem.

  * These are the two empiric antibiotic therapies that every strain is susceptible to.
  * If a patient is allergic to only one of these medications, they may still be approached for enrollment.
* A history of allergy to any of the investigational products/components.
* Patients with liver disease from Hepatitis C.
* Patients with existing inflammatory arthritis.
* History of total colectomy.
* Patients who do not intend to continue their care on a routine basis at the University of Chicago beyond 6 months from the time of enrollment.
* Patients with untreated psychiatric conditions, including illicit substance use disorders, that may interfere with reliable follow-up.
* Unable to participate based on medical judgement of the care team.
* Special populations:

  * Women of childbearing age will have a:

    * Negative serum pregnancy test at screening
    * Use a medically acceptable and highly effective method of birth control for at least 6 weeks following completion of treatment.
  * Another investigational drug or LBP:

    * Prior use will be permitted;
    * Concurrent use will preclude enrollment;
    * Use will be restricted for the duration of the study (12 months after commensal consortia completion)
  * Patients who are prescribed ACE-inhibitors and receive a consortium containing C. comes will receive more frequent blood pressure monitoring.
  * Patients who are prescribed metformin will require either:

    * Switch to another medication for diabetes control; or
    * More frequent Vitamin B12 monitoring at 1, 3, 6, and 12 months of enrollment.
* If a Vitamin B12 deficiency is discovered, it will be repleted as clinically indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2027-08-04 (Estimated); Study Completion 2028-02-04 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events (AEs and SAEs) attributable to the Commensal Consortia | Day 1- Month 12
  Adverse events will be monitored for 1 year after Commensal Consortium administration using in-person contact, telephone calls and/or Patient-Reported Outcomes
Patient-Reported Outcomes Measurement Information System (PROMIS) scores after Commensal Consortia administration | Day 1- Month 12
  Tolerability will be assessed for 1 year after Commensal Consortium administration through completion of PROMIS surveys.
  Surveys will be obtained by the investigators using in-person contact, telephone calls and/or Patient-Reported Outcomes.

SECONDARY OUTCOMES:
The presence of administered bacterial strains in fecal samples | Day 1- Month 12
  Stool samples will be collected at regular intervals and subjected to shotgun metagenomic sequencing. Strain engraftment will be defined as detection of the administered strains.

OTHER OUTCOMES:
Metabolite concentrations in fecal samples | Day 1- Month 12
  Concentrations of targeted metabolites will be measured in fecal samples collected at regular intervals after Commensal Consortium administration.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No